CLINICAL TRIAL: NCT04414475
Title: A Phase 2b, Open-label, Multi-arm Clinical Trial of Selinexor Plus Low-dose Dexamethasone (Sd) in Patients With Penta-refractory Multiple Myeloma or Selinexor and Bortezomib Plus Low-dose Dexamethasone (SVd) in Patients With Triple-class Refractory Multiple Myeloma
Brief Title: A Study of Selinexor (Seli) + Low-dose Dexamethasone (LDD) in Penta-refractory Multiple Myeloma (MM), Seli and Bortezomib + LDD in Triple-class Refractory MM.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XPORT-MM-028
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma, Refractory
Keywords: Multiple Myeloma; Selinexor; Penta-refractory Multiple Myeloma; Triple-class Refractory Multiple Myeloma; KPT-330
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; Dexamethasone; Calcium Dobesilate; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Selinexor + Low-dose Dexamethasone (Sd-40 BIW) (Experimental): Participants will receive fixed dose of 40 milligram (mg) of Selinexor oral tablet followed by 20 mg of low-dose Dexamethasone oral tablet twice weekly (BIW) on Days 1, 3, 8, 10, 15, 17, 22, and 24 of each 28-day cycle.
  Interventions: Drug: Selinexor; Drug: Dexamethasone
- Selinexor + Low-dose Dexamethasone (Sd-100 QW) (Experimental): Participants will receive fixed dose of 100 mg of Selinexor oral tablet followed by 40 mg of low-dose Dexamethasone oral tablet once weekly (QW) on Days 1, 8, 15, and 22 of each 28-day cycle. (Dexamethasone may be given as 20 mg on days 1 and 2 of each week at the discretion of the treating physician).
  Interventions: Drug: Selinexor; Drug: Dexamethasone
- Selinexor + Low-dose Dexamethasone (Sd-80 BIW) (Experimental): Participants will receive fixed dose of 80 mg of Selinexor oral tablet followed by 20 mg of low-dose Dexamethasone oral tablet BIW on Days 1, 3, 8, 10,15, 17, 22, and 24 of each 28-day cycle. Closed for recruitment.
  Interventions: Drug: Selinexor; Drug: Dexamethasone
- Selinexor + Bortezomib + Dexamethasone (SVd) (Experimental): Participants will receive fixed dose of 100 mg of Selinexor oral tablet on Days 1, 8, 15, 22, and 29 followed by 1.3 milligram per square-meter (mg/m^2) of Bortezomib subcutaneous (SC) injection on Days 1, 8, 15, and 22 and followed by 40 mg of low-dose Dexamethasone oral tablet on Days 1, 8, 15, 22, and 29 of each 35-day cycle (Dexamethasone dose may be split to 20 mg on days 1 and 2 of each week at the discretion of the treating physician). Closed for recruitment.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Selinexor — Participants will receive Selinexor oral tablets.
  Other Names: KPT-330; XPOVIO
Drug: Dexamethasone — Participants will receive Dexamethasone oral tablets.
  Other Names: Decadron
Drug: Bortezomib — Participants will receive Bortezomib SC injection.
  Other Names: Velcade
  Arms: Selinexor + Bortezomib + Dexamethasone (SVd)

SUMMARY:
The purpose of this study is to assess the efficacy, antitumor activity, safety and tolerability of selinexor plus low-dose dexamethasone in participants with penta-refractory multiple myeloma or selinexor and bortezomib plus low-dose dexamethasone in participants with triple-class refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to (>=)18 years at the time of signing informed consent.
* Written informed consent in accordance with federal, local, and institutional guidelines.
* Measurable MM based on IMWG guidelines as defined by at least one of the following:

  1. Serum M-protein >= 0.5 gram per deciliter (g/dL) by serum protein electrophoresis (SPEP) or, for Immunoglobulin (Ig) A myeloma, by quantitative IgA.
  2. Urinary M-protein excretion >= 200 mg/24 hours.
  3. Free light chain (FLC) >= 100 milligram per liter (mg/L), provided that the FLC ratio is abnormal.
* Only for arms Sd-40 BIW, Sd-100 QW and Sd-80 BIW prior to protocol version (PV) 5.0: Participants must have relapsed or refractory multiple myeloma (RRMM) and have previously received at least 4 anti-MM prior therapies and have MM that is refractory to previous treatment with at least 2 proteasome inhibitors (PIs), at least 2 immunomodulatory agent (IMiDs), and 1 anti-cluster of differentiation (CD38) monoclonal antibody. Refractory is defined as lesser than or equal to (<=) 25 percent (%) response to therapy, or progression during therapy or progression within 60 days after completion of therapy.
* Only for Arms Sd-40 BIW and Sd-100 QW as of PV 5.0: Participants must have RR MM and have been previously treated with >=3 anti-MM therapies (with exposure to at least 2 PI drugs, at least 2 IMiDs, and 1 anti-CD38 monoclonal antibody), and be refractory to at least 1 drug of each class (PI/IMiD/anti-CD38). Refractory is defined as <=25% response to therapy or progression during therapy or progression within 60 days after completion of therapy.
* Only for arm SVd: Participants must have previously received 1 to 5 anti-MM prior therapies and have MM that is refractory to previous treatment with at least 1 PI, at least 1 IMiD, and 1 anti- CD38 monoclonal antibody.
* Eastern Cooperative Oncology Group (ECOG) performance status of <= 2.
* Female participants of childbearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male participants must use an effective barrier method of contraception if sexually active with a female of childbearing potential. For both male and female participants, effective methods of contraception must be used throughout the study and for 7 months for female and 4 months for male following the discontinuation of study treatment.

Exclusion Criteria:

* Active plasma cell leukemia.
* Documented systemic amyloid light chain amyloidosis.
* Active central nervous system MM.
* Only for SVd arm: Greater than Grade 2 peripheral neuropathy or Grade >= 2 peripheral neuropathy with pain at baseline, regardless of whether or not the participant is currently receiving medication.
* Radiation, chemotherapy, immunotherapy, or any other anticancer therapy (including investigational therapies) <= 2 weeks prior to Cycle 1 Day 1 (C1D1). (Steroids are permitted up to 1 pulse of 40 mg per day for 4 days in the 2 weeks prior to C1D1).
* Active graft vs. host disease (after allogeneic stem cell transplantation) at C1D1.
* Ongoing clinically significant non-hematological toxicities from prior treatments that are Grade greater than (>) 2 at C1D1.
* Inadequate hepatic function defined as total bilirubin >= 2x upper limit of normal (ULN) (>= 3x ULN for participants with Gilbert's syndrome), aspartate transaminase (AST) >= 2.5x ULN, and alanine transaminase (ALT) >= 2.5x ULN.
* Inadequate renal function defined as estimated creatinine clearance of lesser than (<) 20 milliliter per minute (mL/min), calculated using the formula of Cockroft and Gault.
* Inadequate hematopoietic function defined as the following:

  1. Absolute neutrophil count (ANC) < 1000/cubic millimeter (mm^3)
  2. Platelet count < 75,000/mm^3
  3. Hemoglobin (Hb) level < 8.5 g/dL
* Life expectancy of < 4 months, based on the opinion of the Investigator.
* Major surgery within 4 weeks prior to C1D1.
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to first dose.
* Active gastrointestinal dysfunction interfering with the ability to swallow tablets, or any gastrointestinal dysfunction that could interfere with absorption of the study treatment.
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus RNA or hepatitis B virus surface antigen.
* Female participants who are pregnant or lactating.
* Known intolerance, hypersensitivity, or contraindication to glucocorticoid therapy at C1D1.
* Concurrent therapy with approved or investigational anticancer therapeutic including topical therapies.
* Prior exposure to a SINE compound, including selinexor.
* Serious, active psychiatric or active medical conditions which, in the opinion of the Investigator or the Sponsor, could interfere with the participation in the study.
* Contraindication to any of the required concomitant drugs or supportive treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From the date of randomization up to death (approximately 60 months)

SECONDARY OUTCOMES:
Duration of Response (DOR) | From the date of randomization to first disease progression or death (approximately 60 months)
Clinical Benefit Rate (CBR) | From the date of randomization up to death (approximately 60 months)
Disease control rate (DCR) | From the date of randomization up to death (approximately 60 months)
Progression-Free Survival (PFS) | From the date of randomization to first disease progression or death (approximately 60 months)
Overall Survival (OS) | From the date of randomization up to death (approximately 60 months)
Time to Next Treatment (TTNT) | From the date of first dose up to death (approximately 60 months)
Number of Participants with Adverse Events (AE) | From start of study drug administration up to follow-up (approximately 60 months)

CONTACTS AND LOCATIONS:
Locations (16):
- Greece (4):
  - University General Hospital of Patras, Pátrai, Achaia
  - General Hospital of Athens "Alexandra", Attiki, Athens
  - General Hospital of Athens "Evangelismos", Athens, Attica
  - Theageneion Cancer Hospital, Thessaloniki, Thessaloniki
- Israel (12):
  - Emek Medical Center, Afula, Afula
  - Assuta Ashdod Medical Center, Ashdod, Ashdod
  - Bnai-Zion Medical Center, Haifa, Haifa District
  - Rambam Health Care Campus, Haifa, Haifa District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rabin Medical Center (Beilinson Hospital), Petah Tikva, Petah Tikva
  - The Chaim Sheba Medical Center at Tel HaShomer, Ramat Gan, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Meir Medical Center, Kfar Saba

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] White D, Schiller GJ, Madan S, Lentzsch S, Chubar E, Lavi N, Van Domelen DR, Bentur OS, Baljevic M. Efficacy and safety of once weekly selinexor 40 mg versus 60 mg with pomalidomide and dexamethasone in relapsed and/or refractory multiple myeloma. Front Oncol. 2024 May 17;14:1352281. doi: 10.3389/fonc.2024.1352281. eCollection 2024. PMID 38826786